CLINICAL TRIAL: NCT02638077
Title: A Multi-center, Prospective Study to Observe the Initial Management of Patients With Differentiated Thyroid Cancer in the Real World in China (DTCC Study)
Brief Title: Initial Management in Patients With Differentiated Thyroid Cancer in the Real World in China
Acronym: DTCC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Collaborators: West China Hospital (Other); First Affiliated Hospital of Kunming Medical University (Other); Sir Run Run Shaw Hospital (Other); Jilin University (Other); Chinese PLA General Hospital (Other); Gansu Cancer Hospital (Other); Tongji Hospital (Other); First Hospital of China Medical University (Other)
Responsible Party: Principal Investigator, Tao Huang, Director of breast and thyroid department of Wuhan Union Hospital, Tongji Medical College, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Other Study IDs: EMR200125_621
Record Dates: First submitted 2015-12-18; First posted 2015-12-22 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-12

CONDITIONS: Differentiated Thyroid Cancer
Keywords: Differentiated Thyroid Cancer; the initial management

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — tumors samples will retained for detecting gene mutation
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Group 1: 2000 DTC patients undergo the first-time thyroidectomy and identified as intermediate or high risk of recurrence will be recruited. Doctors can treat the patients based on disease conditions. Investigators will record data which are related to study endpoints.

SUMMARY:
* To find out the gap between real-world clinical practice and guideline recommendations in initial management of DTC patients
* To observe the characteristics of patients who achieved and did not achieve TSH target value after one year follow-up
* To assess response to initial therapy in patients who undergo total or near-total thyroidectomy and RAI remnant ablation after one year follow-up (according to an modified dynamic risk stratification system)
* To observe the recurrence status after one year follow-up

DETAILED DESCRIPTION:
Multi-center, prospective, registry study

2000 DTC patients undergo the first-time thyroidectomy and identified as intermediate or high risk of recurrence will be recruited. Doctors can treat the patients based on disease conditions. Investigators will record data which are related to study endpoints.

Primary endpoint(s):

1. Proportion of patients who underwent total/near-total thyroidectomy
2. Proportion of patients who were treated by 131I after undergoing total/near-total thyroidectomy
3. Proportion of patients who achieved serum TSH target value
4. Proportion of patients who did not achieve serum TSH target value although they were treated by TSH suppression therapy

Secondary endpoint(s):

1. Time to achieve serum TSH target value
2. Dosage of L-T4 for patients who achieved and did not achieve serum TSH target value
3. Dosage of L-T4 per kilogram of body weight for patients who achieved and did not achieve serum TSH target value
4. Proportion of excellent response/Acceptable response/Biochemical incomplete response/Structural incomplete response to initial management in patients who undergo total or near-total thyroidectomy and RAI remnant ablation after one year follow-up
5. Recurrence rate after one year follow-up
6. AEs related to L-T4 (or thyroid tablet)treatment

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are diagnosed as DTC (the diagnosis should base on pre-operative examinations and post-operative pathology report)
2. Patients who undergo the first-time thyroidectomy
3. Patients who are identified as intermediate-risk or high-risk of recurrence after thyroidectomy (according to the recurrence risk stratification of Chinese management guideline for patients with thyroid nodules and differentiated thyroid cancer published in 2012)
4. Patients who have Chinese nationality
5. Patients who have signed an informed consent form

Exclusion Criteria:

1. History of thyroid surgery
2. Other malignant tumors
3. Severe organ damage such as heart failure of New York Heart Association classes III-IV, liverfailure, respiratory failure, renal failure, etc.
4. Medical or psychological condition that would not permit the patient to complete the study or sign the informed consent
5. Legal incapacity or limited legal capacity
6. Unwilling to be followed up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Differentiated Thyroid Cancer patients undergo the first-time thyroidectomy and identified as intermediate or high risk of recurrence will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who underwent total/near-total thyroidectomy | one year
2. Proportion of patients who were treated by 131I after undergoing total/near-total thyroidectomy | one year
Proportion of patients who achieved serum TSH target value | one year
4. Proportion of patients who did not achieve serum TSH target value although they were treated by TSH suppression therapy | one year

SECONDARY OUTCOMES:
Time to achieve serum TSH target value | one year
Dosage of L-T4 for patients who achieved and did not achieve serum TSH target value | one year
3. Dosage of L-T4 per kilogram of body weight for patients who achieved and did not achieve serum TSH target value | one year
4. Proportion of excellent response/Acceptable response/Biochemical incomplete response/Structural incomplete response to initial management in patients who undergo total or near-total thyroidectomy and RAI remnant ablation after one year follow-up | one year
Recurrence rate after one year follow-up | one year
AEs related to L-T4 (or thyroid tablet)treatment | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
Not yet

REFERENCES:
- [Derived] Li C, Li S, Zhao Y, Zhang D, Fu Y, Zhou L, Li J, Li F, Du R, Liang N, Sun H. Prognostic Value of Hematological Inflammatory Indices (PLR, NLR, SII) in Medium and High-Risk Papillary Thyroid Carcinoma: A Multicenter Cohort Study. Clin Endocrinol (Oxf). 2025 Oct 16. doi: 10.1111/cen.70046. Online ahead of print. PMID 41102848